CLINICAL TRIAL: NCT03359083
Title: Investigation of the Relationship Between Foot-ankle Characteristics and Lumbopelvic Control, Balance and Physical Performance in Healthy Young Adults.
Brief Title: Relationship Between Foot-ankle Characteristics and Lumbopelvic Control, Balance and Physical Performance
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, CKarartı, Hacettepe University
Other Study IDs: 2017200
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Lumbar Spine Instability; Balance; Physical Performance; Foot; Ankle Deformity
Keywords: foot-ankle characteristic; lumbopelvic control; balance; physical performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Correlation — Correlation between assesment parameters

SUMMARY:
It has been shown that foot and ankle postural disorders can alter the biomechanic of lower extremity and pelvis. This situation can affects balance, postural control and phsical performance of individual adversely. However, it is unknown whether the muscles that control lumbopelvic are affected or not affected. The aim of this study is to investigate the relationship between foot-ankle characteristics and lumbopelvic control, balance and physical performance in healthy young adults.

DETAILED DESCRIPTION:
A healthy load distribution at the foot depends on the ability of the foot to fulfill both the task of stabilization and mobilization. Studies related foot movement disorders usually focus on subtalar joint. The reason for this is that subtalar joint transmits the rotations which in leg to the foot. One of the deformities affecting the foot and subtalar joint is pes planus. Kosashvili et al. have shown that grade 2 and 3 pes planus can affect the lower limb biomechanical alignment, resulting in an increase in perceived pain associated with the knee, hip and pelvic region. Problems related to foot and ankle can affect the balance of individuals as well as affect the pelvic region. Sung et al. have shown that the postural stability and balance of individuals with pes planus are worse than those without pes planus. Studies showing that foot-ankle postural disorders negatively affect physical fitness and motor performance of individuals are also present. Akaras et al. have stated that the increase in pronation in the hindfoot affects individuals' leap and agility performance negatively. It has shown that leg-related problems can affect upper. However, there is no objective study of ultrasonographic imaging of core muscles in foot-ankle problems. The aim of this study is to investigate the relationship between foot-ankle characteristics and lumbopelvic control, balance and physical performance in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate.
* Be between the ages of 18 and 25
* Being a normal weighted individual with a body mass index from 18.5 to 24.9

Exclusion Criteria:

* Presence of any systemic, locomotive or foot related problem
* Undergone any surgical operation related to the foot
* To have loss of sense, diabetic or peripheral neuropathy
* The presence of any problem with the spine (back pain, scoliosis, past surgeons)
* Presence of any neurological problem

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 64 healthy young adults
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2017-12-20 (Estimated); Study Completion 2018-01-20 (Estimated)

PRIMARY OUTCOMES:
INVESTIGATION OF THE RELATIONSHIP BETWEEN FOOT-ANKLE CHARACTERISTICS AND LUMBOPELVIC CONTROL, BALANCE AND PHYSICAL PERFORMANCE IN HEALTHY YOUNG ADULTS | 2 months
  Adverse changes in foot-ankle characteristics in healthy young adults affect lumbopelvic control, balance and phsical performance adversely.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Redmond AC, Crane YZ, Menz HB. Normative values for the Foot Posture Index. J Foot Ankle Res. 2008 Jul 31;1(1):6. doi: 10.1186/1757-1146-1-6. PMID 18822155
- [Background] Richardson CA, Snijders CJ, Hides JA, Damen L, Pas MS, Storm J. The relation between the transversus abdominis muscles, sacroiliac joint mechanics, and low back pain. Spine (Phila Pa 1976). 2002 Feb 15;27(4):399-405. doi: 10.1097/00007632-200202150-00015. PMID 11840107
- [Background] Pinto RZ, Souza TR, Trede RG, Kirkwood RN, Figueiredo EM, Fonseca ST. Bilateral and unilateral increases in calcaneal eversion affect pelvic alignment in standing position. Man Ther. 2008 Dec;13(6):513-9. doi: 10.1016/j.math.2007.06.004. Epub 2007 Oct 1. PMID 17910932